CLINICAL TRIAL: NCT00137410
Title: Protocol For A Multicentre, Double Blind, Parallel Group Pilot Study To Compare Celecoxib Long Term Vs Celecoxib Short Term Therapy In Treatment And Prevention Of New Flare In Patients With Osteoarthritis Of The Knee
Brief Title: Celebrex Short Versus Long Therapy In Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Directorm Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 635-IFL-0508-015; A3191091
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2006-07

CONDITIONS: Osteoarthritis,Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

INTERVENTIONS:
Drug: Celebrex

SUMMARY:
This is a phase III, multicentre, randomized, double blind, parallel-group, pilot study designed to compare a long term (12 weeks) versus a short term (2 weeks) treatment with celecoxib 200 mg/die in treatment and prevention of new flare in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of OA of the knee according to the ACR Classification Criteria for osteoarthritis;
* patients in flare

Exclusion Criteria:

* any concomitant inflammatory rheumatic condition which may interfere with the assessment of OA
* clinical or radiological evidence of chondrocalcinosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Time elapsing between the last drug administration and a new flare, if any, occurring within a 12 months FU and proportion pts with a new flare

SECONDARY OUTCOMES:
Flare intensity WOMAC OA index Psycho-affective Index Pt's assessment of OA pain (VAS) Pt's & Physician's global assessment disease severity Incidence of total AEs Incidence of GI AEs: Incidence of changes in: hematology, renal function, liver function

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Italy (14):
  - Pfizer Investigational Site, Rutigliano, BA
  - Pfizer Investigational Site, Arenzano (GE)
  - Pfizer Investigational Site, Cagliari - Monserrato
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Jesi ( AN)
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Potenza
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Venezia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=635-IFL-0508-015&StudyName=Celebrex+Short+Versus+Long+Therapy+In+Ostheoarthritis+Of+The+Knee